CLINICAL TRIAL: NCT01307176
Title: Exercise Training Program for Cerebellar Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amy J. Bastian, Ph.D., Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00008601; 2R01HD040289-05A1 (NIH)
Record Dates: First submitted 2011-02-23; First posted 2011-03-02 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Cerebellar Ataxia
Keywords: ataxia; exercise; training; cerebellar; rehabilitation
MeSH Terms: conditions — Cerebellar Ataxia; Ataxia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home exercise program (Experimental): Balance and walking exercise program
  Interventions: Behavioral: Home exercise program

INTERVENTIONS:
Behavioral: Home exercise program — The home exercise program uses standard physical therapy exercises that have never been rigorously tested for people with cerebellar ataxia. These include sitting balance exercises (e.g. sitting on a peanut-shaped exercise ball and moving arms or legs), standing balance exercises (e.g. weight shifting, moving arms and legs), and walking exercises (e.g. walking heel-to-toe). The exercises are in a progression, going from less to more challenging. Though the exercises are standard, they are the intervention that we are testing and we will consider them experimental.
  Other Names: Woodway Split Belt Treadmill; Company: Woodway USA, Inc

SUMMARY:
The purpose of this study is to determine whether a person's ability to adapt (i.e. short term motor learning) predicts their ability to benefit from physical therapy exercises.

DETAILED DESCRIPTION:
The cerebellum is important for coordination of movement and for motor learning. No medications systematically improve cerebellar ataxia, and little is known about the effectiveness of rehabilitation exercises, which are often the only treatment option. Here, we ask whether a person's ability to adapt (i.e. short term motor learning) predicts their ability to benefit from physical therapy exercises. This pilot-clinical trial will test a subject's ability to adaptively learn a new walking pattern in a single session, and then any improvement of walking and balance over a 13 week time period during which they participate in a specialized home exercise training program. Our prediction is that those individuals with some preserved adaptive learning ability will be the best rehabilitation candidates.

ELIGIBILITY:
Inclusion Criteria:

* Cerebellar damage from stroke, tumor, or degeneration
* Able to stand and take steps with or without assistance
* Age 18-95

Exclusion Criteria:

* Extrapyramidal symptoms
* Peripheral vestibular loss (e.g. absence of VOR)
* Congestive heart failure
* Peripheral artery disease with claudication
* Pulmonary or Renal Failure
* Unstable angina
* Uncontrolled hypertension ( > 190/100 mmHg)
* Dementia (Mini-Mental State exam > 22)
* Severe aphasia
* Orthopedic or pain conditions
* Pregnancy
* Prisoner
* Evidence of chronic white matter disease on MRI

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in walking speed from baseline to mid-training and to post-training | Participants are assessed at baseline (week 1 and week 3), mid-training (week 6), and post-training (week 9 and week 13). There are a total of 13 weeks for this study with 5 visits during that time period
  Here, we ask whether a person's ability to adapt (i.e. short term motor learning) predicts their ability to benefit from physical therapy exercises. Our prediction is that those individuals with some preserved adaptive ability will be show the greatest improvement in walking speed.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Bastian, PhD, PT, Principal Investigator — Kennedy Krieger Institute and Johns Hopkins School of Medicine
Locations (1):
- Motion Analysis Lab in the Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- See also: Motion Analysis Lab website at the Kennedy Krieger Institute — http://www.kennedykrieger.org/kki_research.jsp?pid=5741